CLINICAL TRIAL: NCT03365128
Title: Enhancing Operability in a Hypobaric Hypoxic Environment With a Small Oxygen Storage System
Status: Withdrawn | Type: Observational
Why Stopped: Could not obtain regulatory approval
Sponsor: University of Cincinnati (Other)
Responsible Party: Principal Investigator, Chris Blakeman, Instructor, University of Cincinnati
Other Study IDs: Blakeman2017
Record Dates: First submitted 2017-12-01; First posted 2017-12-07 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Hypobaric Hypoxemia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This is a study to validate the efficacy of using a small portable oxygen source to mitigate altitude-induced hypoxia.

DETAILED DESCRIPTION:
The purpose of this study is to validate the efficacy of using a small portable oxygen source to mitigate altitude-induced hypoxic events. To do so, the invesitgators propose the following aims:

1. Determine the ability of a portable oxygen storage device to reverse hypobaric hypoxemia in volunteers at altitude.
2. Determine the duration of time that a single portable oxygen container can maintain normoxia in normal volunteers at altitude.
3. Determine the optimum dose and timing of oxygen use to reverse hypobaric hypoxemia.

ELIGIBILITY:
Inclusion Criteria:

* Altitude chamber qualified
* Previous agreement to be approached regarding altitude chamber research

Exclusion Criteria:

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Normal volunteers aged 18 to 65 years, inclusive
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2025-05-28 (Actual); Study Completion 2025-05-28 (Actual)

PRIMARY OUTCOMES:
Elapsed time during which oxygen saturation by pulse oximetry (SpO2) remains above 90% I | 15 minutes
  Elapsed time during which subject's SpO2 remains above 90% after initially reaching or exceeding 94% following exposure to a simulated altitude of 14,000 and after receiving pulse-dosed oxygen

SECONDARY OUTCOMES:
Amount of oxygen needed to return SpO2 to sea level value I | 15 minutes
  Amount of oxygen needed to return subject's SpO2 value to 94% (or higher) after exposure to a simulated altitude of 14,000 feet
Amount of oxygen needed to return SpO2 to sea level value II | 15 minutes
  Amount of oxygen needed to return subject's SpO2 value to 94% (or higher) after (i) reaching SpO2 value of 82-84% or (ii) attaining 85% of maximum predicted heart rate. This is following exercise on a stationary bicycle at a simulated altitude of 10,000 feet
Elapsed time during which SpO2 remains above 90% II | 15 minutes
  Elapsed time during which subject's SpO2 remains above 90% after initially following exposure to a simulated altitude of 14,000 and after initially (i) reaching SpO2 value of 82-84% or (ii) attaining 85% of maximum predicted heart rate. This is following exercise on a stationary bicycle at a simulated altitude of 10,000 feet and after receiving pulse-dosed oxygen.

IPD SHARING:
Plan to Share IPD: No